CLINICAL TRIAL: NCT00602693
Title: Phase I Study of Infusion of Umbilical Cord Blood (UCB) Derived CD25+CD4+ T-Regulatory (Treg) Cells After Nonmyeloablative Cord Blood Transplantation
Brief Title: T-Regulatory Cell Infusion Post Umbilical Cord Blood Transplant in Patients With Advanced Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007LS022; MT2006-01 (Other: Blood and Marrow Transplantation Program); 0701M00303 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-01-10; First posted 2008-01-28 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma; Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: chronic myelogenous leukemia; recurrent mantle cell lymphoma; prolymphocytic leukemia; advanced chronic lymphocytic leukemia; small lymphocytic lymphoma; B-cell lymphoma; follicular lymphoma; diffuse large cell lymphoma; anaplastic large cell lymphoma; Hodgkin lymphoma; multiple myeloma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Mantle-Cell; Leukemia, Prolymphocytic; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic; Hodgkin Disease | interventions — Cord Blood Stem Cell Transplantation; Allopurinol; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Radiation; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UCB post-transplant Treg Cell Infusion (Experimental): Includes patients with high risk malignancy receiving allopurinol, fludarabine phosphate, cyclophosphamide, sirolimus, total body irradiation, double umbilical cord blood transplantation and Treg infusion cells after transplant. Patients will receive differing dose levels as they are entered and assigned to determine the maximum tolerated dose.
  Interventions: Biological: umbilical cord blood transplantation; Drug: Allopurinol; Drug: fludarabine phosphate; Drug: Cyclophosphamide; Radiation: Total body irradiation; Biological: Treg infusion; Drug: Sirolimus

INTERVENTIONS:
Biological: umbilical cord blood transplantation — Infusion of umbilical cord blood
  Other Names: UCB transplant
Drug: Allopurinol — Administration begins Day -7 through Day 0, tablet or powder prescribed on an individual basis.
  Other Names: Zyloprim
Drug: fludarabine phosphate — 40 mg/m^2 intravenously over 1 hour on Days -6, -5, -4, -3, -2
  Other Names: Fludara
Drug: Cyclophosphamide — 50 mg/kg intravenous over 2 hours on Day -6
  Other Names: Cytoxan
Radiation: Total body irradiation — 200 cGy on Day -1
  Other Names: radiation
Biological: Treg infusion — Infusion of T regulatory cells on Day +1 (also Day +15 for Dose level 5 only). Dose escalation ranges include 1, 3, 10, 30, 100, 300 1000, and 300 x 10^5 Treg/kg.
  Other Names: Treg cells
Drug: Sirolimus — Beginning on day -3 and continuing until day +100, patients receive sirolimus intravenously (IV) with 8-12 mg oral loading dose followed by a single dose of 4mg/day with a target serum concentration of 3-12 mg/mL with a taper until day +180.
  Other Names: Rapamune®

SUMMARY:
RATIONALE: Giving chemotherapy, such as fludarabine and cyclophosphamide, and total-body irradiation before a donor umbilical cord blood transplant helps stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T-regulatory cells after the transplant may decrease this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. However, the donor immune system may also react against the recipient's tissues (graft-versus-host disease).

PURPOSE: This phase I trial is studying the side effects and best dose of donor T-regulatory cells after an umbilical cord blood transplant in treating patients with advanced hematologic cancer or other disorder.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of umbilical cord blood (UCB)-derived T-regulatory (Treg) cells.

Secondary

* Estimate the proportion of patients with detectable circulating Treg cells at 0, 1, 3, 7, and 14 days after infusion.
* Estimate the risk of grades II-IV and III-IV acute graft versus host disease (GVHD) at day +100 with the infusion of Treg cells.
* Estimate the proportion of patients with sustained donor engraftment.
* Estimate the proportion of patients with double chimerism at 6 months and 1 year.
* Determine the speed and cumulative incidence of neutrophil recovery by day 42 and platelet recovery by 6 months after UCB transplantation.
* Estimate the risk of chronic GVHD at 1 year.
* Estimate the probability of disease-free survival at 100 days and 1 year.
* Estimate the risk of fungal and viral infections at 1 year
* Estimate the risk of relapse at 1 year
* Characterize the pattern of immune cell recovery over 1 year

OUTLINE: This is a dose-escalation study of umbilical cord blood (UCB)-derived T-regulatory (Treg) cells. Patients receive nonmyeloablative UCB transplantation and post-transplant immunosuppression as in protocol UMN-2005LS036 (without antithymocyte globulin during conditioning regimen).

* Nonmyeloablative conditioning and UCB transplantation: Patients receive allopurinol on days -7 to day 0, fludarabine phosphate intravenously (IV) over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on day -6; undergo total-body irradiation (TBI) once on day -1; and undergo UCB transplantation on day 0.
* Immunosuppression therapy: Beginning on day -3 and continuing until day +100, patients receive sirolimus intravenously (IV) with 8-12 mg oral loading dose followed by a single dose of 4mg/day with a target serum concentration of 3-12 mg/mL with a taper until day +180. Patients also receive mycophenolate mofetil IV or orally every 8 hours on days -3 to +30.
* Radiation therapy: total body irradiation is administered on Day -1 of 200 cGy.
* UCB Treg cell infusion: Patients receive escalating doses of UCB-derived CD4+ CD25+ Treg cells IV on day +1 (and Day +15 for dose level 5 only) until the maximum tolerated dose is obtained.

After completion of study treatment, patients are followed at day 180, 360, and 720.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 75 years old
* Eligible for and co-enrolled on protocol UMN-2005LS036, for treatment of any of the following advanced hematologic malignancies:

  * Acute leukemias in complete remission (high risk CR1 or subsequent CR); chronic myelogenous leukemia (except refractory blast crisis); myelodysplastic syndrome with severe pancytopenia or complex cytogenetics, large-cell lymphoma, Hodgkin's lymphoma and multiple myeloma, chronic lymphocytic leukemia/small lymphocytic lymphoma, marginal zone b-cell lymphoma, follicular lymphoma, lymphoplasmacytic lymphoma, mantle-cell lymphoma, prolymphocytic leukemia may be eligible after initial therapy.
* Have three partially HLA matched umbilical cord blood (UCB) units (1-2 units for UCB transplantation per MT2005-02 and 1 unit for the Treg cell infusion.)
* Adequate organ function

Exclusion Criteria:

* Patients not exposed to highly immunosuppressive single agent or multi-agent chemotherapy within 3 months, or an ablative preparative regimen for autologous hematopoietic stem cell transplant (HCT) within 1 year.
* Pregnancy or breastfeeding
* Current active serious infection
* Evidence of human immunodeficiency virus (HIV) or known HIV positive serology
* Patients with acute leukemia in morphologic relapse/persistent disease defined as >5% blasts in a > or = 15% cellular bone marrow or any % blasts if blasts have unique morphologic markers (e.g., Auer rods) or associated cytogenetic markers that allows morphologic relapse to be distinguished are not eligible.
* Chronic myelogenous leukemia in refractory blast crisis.
* Active central nervous system malignancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-07-23 (Actual); Primary Completion 2014-09-25 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 48 Hours
  Nine dose levels of CD4+CD25+ Treg are scheduled with the doses being 1, 3, 10, 30, 30+30, 100, 300, 1000, and 3000 x 10^5 Treg/kg recipient body weight. The dose escalation will proceed in cohorts of one patient until the first dose limiting toxicity (DLT) is observed.

SECONDARY OUTCOMES:
Number of patients with detectable Treg cells | Days 0, +1, +3, +7, and +14 after Treg cell infusion
  determined by polymerase chain reaction (PCR) and flow cytometry
Number of Patients with grade II-IV and grade III-IV acute graft versus host disease (GVHD) | Day 100
  Patients will be assessed weekly for GVHD between days 0 and 100 after transplantation using standard criteria. Patients will be assigned an overall GVHD score based on extent of skin rash, volume of diarrhea and maximum bilirubin level. Incidence of grades II-IV and grades III-IV GVHD by day 100 will be monitored.
Number of patients with sustained donor engraftment | Day 100
Number of patients with double chimerism | 6 Months and 1 Year
Incidence of neutrophil recovery after umbilical cord blood (UCB) transplantation | Day 42
Number of Patients with Chronic Graft Versus Host Disease (GVHD) | 1 Year
Number of Patients with disease-free survival | Day 100 and 1 Year
Number of Patients with Fungal and Viral Infections | 1 Year
  Count of reported infections.
Incidence of platelet recovery after umbilical cord blood (UCB) | 6 Months After Transplant
Number of Patients with Disease Relapse | 1 Year
Percent of Patients with Immune Cell Recovery | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Claudio G. Brunstein, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota; Margaret L. MacMillan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Brunstein CG, Miller JS, Cao Q, McKenna DH, Hippen KL, Curtsinger J, Defor T, Levine BL, June CH, Rubinstein P, McGlave PB, Blazar BR, Wagner JE. Infusion of ex vivo expanded T regulatory cells in adults transplanted with umbilical cord blood: safety profile and detection kinetics. Blood. 2011 Jan 20;117(3):1061-70. doi: 10.1182/blood-2010-07-293795. Epub 2010 Oct 15. PMID 20952687